CLINICAL TRIAL: NCT04108780
Title: Comparative Study : Repair of Common Bile Duct After CBD Exploration Over T-tube or Primary Repair Without Tube
Brief Title: CBD Repair Over T-tube or Primary Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Aboelhassan Mohamed Hassanein, doctor, Assiut University
Other Study IDs: CBD exploration
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: CBD Exploration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CBD exploration with T-tube: repair of CBD after CBD exploration over T-tube
  Interventions: Device: T-tube
- CBD exploration with primary repair: primary repair of CBD after CBD exploration
  Interventions: Device: T-tube

INTERVENTIONS:
Device: T-tube — T shaped tube used as stent after CBD exploration

SUMMARY:
the aim is to assess the benefits and harms of T-tube drainage versus primary closure without biliary stent after exploration common bile duct stones

DETAILED DESCRIPTION:
Common Bile Duct Exploration is a surgery that involves opening the main bile duct that drains from liver and gallbladder into the first part of the small intestine (the duodenum). This is needed when a gallstone drops out of the gallbladder into the duct and partially or completely blocks up the duct. This can cause jaundice , fever and chills, severe abdominal pain due to infection / inflammation of the bile duct, gallbladder or pancreas. This most often involves admission to the hospital and urgent intervention. Most commonly, a procedure called an ERCP is used to clear out the stones from the bile duct. If gallbladder will have to be removed soon to prevent this potentially serious condition from occurring again.

During the operation the investigators remove gallbladder then a duct exploration is performed. This involves opening the duct directly and removing the stones.

Prior to Common Bile Duct Exploration surgery, patient will be asked not to eat anything after midnight prior to the surgery. patient will be given specific instructions from the surgeon or anesthesiologist about which medications he should or should not take prior to the surgery. patient should not take any blood thinning medications at least 5 days prior to your operation. This should be discussed with the surgeon at the preop visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo common bile duct exploration

Exclusion Criteria:

* patients who has failed ERCP for management of common bile duct exploration
* CBD diameter 2 cm or more

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patient who will undergo CBD exploration for management of CBD stone
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-25 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
bile leak from common bile duct | baseline
  Assessment which type of repair (with T-tube or primary repair) bile leak will occurs more

SECONDARY OUTCOMES:
hospital stay length | base line
  Assessment which type of repair (with T-tube or primary repair) patient will stay in the hospital more after CBD exploration

REFERENCES:
- [Background] Wu X, Huang ZJ, Zhong JY, Ran YH, Ma ML, Zhang HW. Laparoscopic common bile duct exploration with primary closure is safe for management of choledocholithiasis in elderly patients. Hepatobiliary Pancreat Dis Int. 2019 Dec;18(6):557-561. doi: 10.1016/j.hbpd.2019.07.005. Epub 2019 Jul 25. PMID 31474445
- [Background] Guan H, Jiang G, Mao X. Primary duct closure combined with transcystic drainage versus T-tube drainage after laparoscopic choledochotomy. ANZ J Surg. 2019 Jul;89(7-8):885-888. doi: 10.1111/ans.15163. Epub 2019 May 8. PMID 31067598
- [Background] Jiang C, Zhao X, Cheng S. T-Tube Use After Laparoscopic Common Bile Duct Exploration. JSLS. 2019 Jan-Mar;23(1):e2018.00077. doi: 10.4293/JSLS.2018.00077. PMID 30675097